CLINICAL TRIAL: NCT06456983
Title: Maintenance ElectroConvulsive Therapy in Clozapine RESISTant Schizophrenia - the MECT-RESIST Trial
Acronym: MECT-RESIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MECT-RESIST; 01KG2401 (Other Grant/Funding Number: Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2024-01-30; First posted 2024-06-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia; Treatment Resistant Schizophrenia
Keywords: electroconvulsive therapy; ECT
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: This is a multi-center, observer-blind, randomized, and actively controlled parallel-group clinical trial to examine the effectiveness of mECT in clozapine resistant patients with schizophrenia (CRS) who improved after a full course of routine ECT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment as usual (TAU) (No Intervention): Patients randomized to TAU only will continue on a stable drug regime for the next 28 weeks, but will not receive maintenance electroconvulsive therapy (mECT)
- maintenance electroconvulsive therapy (mECT) plus TAU (Active Comparator): All subjects will enter PHASE 1 and will receive a full course of routine ECT (maximum of 9 weeks and 18 total ECTs with 2-3 treatments per week) while being on stable antipsychotic medication. All ECT-responders (patients with improvement of 30% or more on Brief Psychiatric Rating Scale (BPRS) will enter PHASE 2 and will be randomly assigned to the active comparator (mECT plus treatment-as-usual, TAU) or the control intervention (TAU) which both last 28 weeks. Non-responders (patients without improvement of at least 30 % on BPRS scale) will not enter PHASE 2.
  Interventions: Device: maintenance electroconvulsive therapy (mECT)

INTERVENTIONS:
Device: maintenance electroconvulsive therapy (mECT) — see Arms
  Arms: maintenance electroconvulsive therapy (mECT) plus TAU

SUMMARY:
Schizophrenia is one of the most severe and costliest mental disorders in terms of human suffering and societal expenditure. About 15-30% of patients do not respond to all known antipsychotics, including clozapine, the current gold-standard in these cases. Hence, a recent Cochrane review stated that the quality of the existing studies is too poor to recommend any intervention in addition to clozapine and that new, randomized controlled trials independent from the pharmaceutical industry need to be performed to substantially improve patient care. Although electroconvulsive therapy (ECT) was initially used to treat schizophrenia, it is nowadays by far underused in the therapy of schizophrenia in many countries. ECT is well known to be highly effective in clozapine-treatment-resistant schizophrenia (CRS), and synergistic effects of clozapine and ECT have been demonstrated. However, relapse rates after successful courses of ECT are still very high, and evidence for maintenance ECT (mECT) in CRS is scarce at best. In a multi-center trial the investigators aim to examine the effectiveness of mECT in treatment-resistant patients with schizophrenia who improved after a course of routine ECT. If mECT will lead to a later timepoint of relapse and/or to a higher proportion of relapse-free patients compared to those undergoing treatment as usual, this trial would have an enormous impact on therapeutic strategies for "treatment-resistant" patients and would induce a profound change of current treatment guidelines, where ECT still ranks at the level of ultima ratio, despite accumulating evidence suggesting otherwise.

DETAILED DESCRIPTION:
The scientific aim of the study is to conduct a multicenter, blinded, randomized and actively controlled trial to test the hypothesis that maintenance ECT (mECT) plus clozapine is superior to treatment with clozapine alone in CRS. Prior to the start of mECT (phase II), an acute ECT series (phase I) should have already led to a significant clinical improvement in CRS patients. The superiority of mECT will be proven by a longer time to relapse and secondarily by a lower number of patients with relapse compared to the control group.

Secondary objectives are to test the hypotheses that the global level of functioning and quality of life will increase, and that depression, overall symptoms of the schizophrenic syndrome, concomitant catatonic symptoms, stress and self-stigmatization will decrease compared to the control group. It is also expected that cognitive performance will not only not deteriorate, but will improve over the course of the mECT.

Once the positive ethics votes have been obtained, the first patients will be included at the individual centers following successful center initiation. In month 12 at the latest, the first patient should leave phase I after 6-9 weeks as a responder and will be randomized in phase II (clozapine versus clozapine plus mECT). At month 30 the last patient (total n = 84) should have been randomized as a responder from phase I and been included in phase II. At month 36 the last planned patient completes phase II of the study with his/her last study visit. Accordingly, he/she is the last patient to start the 12-month follow-up phase. In month 46 investigators will start final data evaluation and analysis. Investigators will complete the primary publication of the study this time point. After 4 years the last patient completes the 12-month follow-up phase. At study end final data evaluation and analysis regarding the primary endpoint of the follow-up phase takes place as well as the completion and submission of the primary publication of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), BPRS total score > 45 and history of clozapine resistant schizophrenia (CRS), which will include treatment-resistant schizophrenia with clozapine intolerance or absolute contraindications for clozapine;

Exclusion Criteria:

1. Diagnosis of DSM-5 major neurocognitive disorder ("dementia"), current severe substance-use disorder, affective disorders with psychotic symptoms or any personality disorder;
2. Inability to read/write German
3. Pregnancy or breast-feeding;
4. General medical condition contraindicating ECT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Time to relapse | 28 weeks (duration of PHASE 2)
  Time to relapse (relapse defined as BPRS 20 % higher than individual BPRS at start of PHASE 2 at any following study visit OR any unscheduled readmission due to a worsening of psychiatric symptoms OR any unscheduled visit with an BPRS 20 % higher than individual BPRS at start of PHASE 2 or death).

SECONDARY OUTCOMES:
Number of relapse free subjects | after 28 weeks, i.e. end of Phase 2
  Number of relapse free subjects at the end of PHASE 2
BPRS | after 28 weeks, i.e. end of Phase 2
  BPRS: Brief Psychiatric Rating scale; higher is worse
GAF: | after 28 weeks, i.e. end of Phase 2
  GAF: Global Assessment of Functioning; higher is better
SLSSWB: | after 28 weeks, i.e. end of Phase 2
  SLSSWB: self-labeling, stigma stress and well-being (SLSSWB); descriptive subscales
PANSS: | after 28 weeks, i.e. end of Phase 2
  PANSS: Positive and Negative Syndrome Scale; higher is worse
HAMD: | after 28 weeks, i.e. end of Phase 2
  HAMD: Hamilton Depression scale; higher is worse
  SSMIS-SF: Self-Stigma of Mental Illness Scale - Short Form; descriptive subscales
NCRS-dv: | after 28 weeks, i.e. end of Phase 2
  NCRS-dv: Northoff catatonia rating scale (German version); higher is worse
Q-LES-Q-18: | after 28 weeks, i.e. end of Phase 2
  Q-LES-Q-18: Quality of Life Enjoyment and Satisfaction Questionnaire (for patients with schizophrenia); higher is better

OTHER OUTCOMES:
Cognition: MMSE: | after 28 weeks, i.e. end of Phase 2
  MMSE: Mini Mental State Examination; higher is better
THINC-it: | after 28 weeks, i.e. end of Phase 2
  THINC-it: Tool for Cognitive Assessment and Measurement; green - amber - red (red means lower than 1 standard deviation worse than healthy control subjects)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sartorius, Prof, Principal Investigator — Central Institute of Mental Health (CIMH), Mannheim, Germany
Locations (14):
- Germany (14):
  - Dept. of Psychiatry, RWTU Aachen, Aachen
  - Dept. of Psychiatry, University of Augsburg, Augsburg
  - Klinik für Psychiatrie, Göppingen, Göppingen
  - Departmet of Psychiatry, University Medical Center Göttingen, Göttingen
  - Dept. of Psychiatry, Hannover Medical School, Hanover
  - Universitätsklinikum Heidelberg, Klinik für Allgemeine Psychiatrie, Heidelberg
  - Zentrum für Psychische Gesundheit, Ingolstadt
  - Dept. of Psychiatry, University Mainz, Mainz
  - Department of Psychiatry and Psychotherapy, Central Institute of Mental Health (CIMH), Mannheim
  - Dept. of Psychiatry, LMU München, München
  - Clinic for Psychiatry, Saarbrücken, Saarbrücken
  - Klinik für Psychiatrie, Siegen, Siegen
  - Dept. of Psychiatry, University Tübingen, Tübingen
  - Dept. of Psychiatry I, Wiesloch, Wiesloch

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deicher A, Karl S, Otte ML, Knabbe J, Wendel B, Gose M, Wolf RC, Sartorius A. Study protocol of a German multi-center, observer-blind, randomized, and actively controlled parallel-group trial comparing maintenance electroconvulsive therapy to treatment as usual for relapse prevention in clozapine resistant schizophrenia. BMC Psychiatry. 2025 May 26;25(1):536. doi: 10.1186/s12888-025-06990-2. PMID 40420043